CLINICAL TRIAL: NCT06895395
Title: High and Low Intensity Speech Intervention in Children With a Cleft Palate: Perceptions of Children, Their Caregivers and Speech-language Pathologists
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Organization: University Hospital, Ghent (Other)
Other Study IDs: ONZ-2024-0191
Record Dates: First submitted 2024-11-27; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cleft Lip and Palate; Speech Disorders in Children
Keywords: Cleft lip and palate; Qualitative research; Speech therapy; Interviews; Speech intervention intensity
MeSH Terms: conditions — Cleft Lip; Communication Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Behavioral: High intensive combined phonetic-phonological intervention — High intensity speech intervention 5 times 30' per week for 2 times 4 weeks
Behavioral: Low intensive combined phonetic-phonological intervention — low intensity speech intervention 2 times 30' per week for 20 weeks

SUMMARY:
A cleft (lip and) palate (CP±L) is the most common congenital abnormality of the face and skull with a significant social impact, affecting speech, hearing, feeding, oral behavior, dentition and satisfaction with appearance. These consequences have a long-term and negative impact on social integration and well-being. The World Health Organization (WHO) highlights the significant financial costs, including morbidity, health care costs, emotional distress and social exclusion for patients, their families and society. The purpose of this study is to compare high- and low-intensity speech intervention in children with CP±L based on the perceptions of the providers of the intervention (primary care speech-language pathologists) and the recipients of the intervention (children with CP±L and their caregivers). Individual semi-structured interviews will be conducted with both intervention providers and recipients to explore perceptions and experiences, as well as acceptability of the two speech intervention intensities. Potential participants will be told that the interview will be recorded. The actual interviews will take place at a location and time that is most convenient for the participants. Each interview will be recorded using a Roland R-05 high-quality audio recorder. After conducting the interviews, all participants will be asked to complete a questionnaire regarding their demographics. In addition, data regarding the type of cleft, time and manner of closure of the cleft, any secondary surgery and otological/audiological data will be collected from the medical records of the children with CP±L. Based on this qualitative study, possible adjustments to the high-intensity therapy protocol can be made. In doing so, these modifications will be relevant to these key stakeholders. This will also facilitate the implementation and widespread use of high-intensity speech therapy in clinical speech therapy practice.

ELIGIBILITY:
Inclusion Criteria:

* Belgian Dutch-speaking children with a cleft palate with or without a cleft lip
* Aged between 4 and 12 years,
* Presence of at least one compensatory speech error in their speech based on the perceptual assessment of one experienced speech-language pathologist

Exclusion Criteria:

* Children with syndromic clefts
* Oronasal fistula
* Velopharyngeal insufficiency
* Hearing disabilities based on pure tone audiometry (>25 dB HL)
* Cognitive and/or related learning disabilities or neuromuscular disorders

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population are children born with a cleft palate (with or without a cleft lip). They are 4 to 12 years old and have at least one compensatory speech error in their speech.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Perceptions and acceptability of low/high intensive speech intervention | 20 weeks
  Participants will be interviewed and can talk about their experiences and perceptions regarding the speech intervention intensity. The acceptability of both high and low intensive therapy will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No